CLINICAL TRIAL: NCT05438082
Title: Antibiotic Prophylaxis to Prevent Post-procedure Urinary Tract Infection After Voiding Cystourethrogram
Brief Title: Antibiotic Prophylaxis to Prevent Post-procedure UTI After VCUG
Acronym: APPrUV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Sarah Khan, Associate Professor, Hamilton Health Sciences Corporation
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19481
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Antibiotic Prophylaxis; Voiding Cystourethrogram; Febrile Urinary Tract Infection
MeSH Terms: interventions — Antibiotic Prophylaxis

STUDY DESIGN:
Intervention Model Description: This trial is a single center, parallel, blinded, randomized, placebo-controlled pilot trial in children
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic Prophylaxis (Experimental): one dose of either Trimethoprim (if < 2 months) or Trimethoprim-Sulfamethoxazole (if ≥ 2 months) or placebo in suspension. Dosing regimen for the active treatment (Trimethoprim) will be based on weight (5mg/kg of Trimethoprim component) with a maximum dosage of 320mg.
  Interventions: Drug: Antibiotic Prophylaxis
- Placebo (Placebo Comparator): The placebo group will receive an equal volume of placebo suspension that has been developed to have the same colour and taste as the antibiotic to preserve blinding.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Antibiotic Prophylaxis — This trial will contain two arms in which patients will be randomized to receive one dose of either Trimethoprim (if < 2 months) or Trimethoprim-Sulfamethoxazole (if ≥ 2 months) or placebo in suspension. Dosing regimen for the active treatment (Trimethoprim) will be based on weight (5mg/kg of Trimethoprim component) with a maximum dosage of 320mg
  Arms: Antibiotic Prophylaxis
Other: Placebo — The placebo group will receive an equal volume of placebo suspension that has been developed to have the same colour and taste as the antibiotic to preserve blinding.
  Arms: Placebo

SUMMARY:
The current practice of pre-VCUG antibiotic prophylaxis is highly variable. A recent unpublished survey of Society of Fetal Urologists (SFU) completed by this study team found that 87% of respondents reported having patients who develop fUTI following VCUG, with 30% of respondents prophylaxing for fUTI in patients undergoing VCUG. The current lack of best practice guidelines regarding antibiotic prophylaxis prior to VCUG due to low quality of current literature, and a growing concern around risks of unnecessary antibiotic exposure suggests the need for an RCT. The results of this pilot trial will inform the ability to conduct a definitive RCT on this important subject. The results of the definitive trial would have important clinical and economic implications.

DETAILED DESCRIPTION:
What are the Study Objectives? The primary objective of this pilot trial is to determine the feasibility of conducting a definitive trial investigating whether pre-VCUG antibiotic prophylaxis, when compared to placebo, decreases the risk of fUTI in infants undergoing VCUG for genitourinary abnormalities. The pilot trial will address specific feasibility outcomes including process, resources, management and scientific domains. The pilot will lay the groundwork for the eventual full trial. Funding for the full trial will be sought after preliminary data is collected from the pilot study.

The primary objective for the definitive trial is to determine whether single-dose, preprocedural antibiotic prophylaxis compared to placebo lowers the risk of fUTI in children < 3 years of age who are undergoing VCUG for the following indications: high-grade (SFU Classification III, IV/UTD 2,3) HN, ureteral dilatation, or bladder abnormalities found during renal ultrasound. The secondary outcomes of the definitive trial will include assessment of adverse event outcomes related to antibiotic prophylaxis administration, including antibiotic resistant UTI pathogens, episodes of antibiotic associated diarrhea, and C. difficile.

ELIGIBILITY:
Inclusion Criteria:

1. Children <3 years of age undergoing VCUG for the following indications: high-grade SFU/UTD hydronephrosis, ureteral dilatation, or bladder abnormalities found during renal ultrasound
2. Parent or legal guardian able to provide informed consent

Exclusion Criteria:

1. Chronic antibiotic use
2. Allergy to Trimethoprim or Trimethoprim-Sulfamethoxazole

Max Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of pilot study: randomization, compliance, enrollment targets | 12 months
  The primary feasibility outcomes for the pilot study will be recruitment rate (>50% of eligible infants enrolled), randomization rate (percentage of participants randomized, >95%), medication compliance rate (>80%), percentage of the primary endpoints (febrile UTI) and cost of being in the trial per patient. We would also aim to demonstrate a <15% rate of protocol violations, and loss to follow-up. The major clinical outcome for the pilot study is to determine the event rate of UTI in patient post-procedure to inform the sample size calculation for the larger trial.

SECONDARY OUTCOMES:
Resource Allocation | 12 months
  Secondary outcomes in the pilot study will be adequacy of research resource allocation, to understand if further study supports are required for the eventual multi-centre trial. Management outcomes include determining research coordinator capacity, processing times for each enrollment, and follow-up, time required for adjudication UTI events, and ensuring adequacy and accuracy of data management. We will also aim to understand potential barriers to recruitment, and compliance. Adverse events related to antibiotic use for patients will be recorded as well.
Febrile UTI within 7 days of VCUG Procedure | 7 days
  Patients will be enrolled in the study for 7 days post VCUG, which is clinically considered the immediate post-procedure period.

IPD SHARING:
Plan to Share IPD: No